CLINICAL TRIAL: NCT03596307
Title: The Effects of Ashwagandha In Endurance Exercise Performance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Arjuna Natural Limited (Industry)
Collaborators: KU Leuven (Other); ZB Sports Development BVBA (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: AN-07SHO 0518H1-ULE02
Record Dates: First submitted 2018-06-28; First posted 2018-07-23 (Actual); Last update posted 2018-11-26 (Actual); Status verified 2018-11

CONDITIONS: Healthy
Keywords: Ashwagandha; Endurance; VO2 max; Glycowithanolides; Shoden
MeSH Terms: interventions — Ashwagandha

STUDY DESIGN:
Intervention Model Description: Randomization 1:1. Acute phase study - Session 1 (2 days) ; Crossover; Session 2 ( 2 Days) Short Term Phase - Session 2 (Pretest), 16 day supplementation, Session 3 (Post test), Crossover; Session 4 (Pretest),16 day supplementation, Session 5 (Post test).
Who Masked: Participant, Investigator
Masking Description: Double blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ashwagandha extract (Experimental): 180 mg Shoden once daily before breakfast for 2 days in Acute Phase and 16 days in Short Term Phase.
  Interventions: Dietary Supplement: Ashwagandha extract; Dietary Supplement: Placebo
- Placebo (Placebo Comparator): 180 mg identical placebo once daily before breakfast for 2 days in Acute Phase and 16 days in Short Term Phase.
  Interventions: Dietary Supplement: Ashwagandha extract; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Ashwagandha extract — Shoden 180 mg capsule.
  Other Names: Shoden; Withania somnifera extract
Dietary Supplement: Placebo — Placebo 180 mg (Sucrose) capsule.

SUMMARY:
Ashwagandha (Withania Somnifera) is a widely used herb in Ayurvedic medicine for vitality and rejuvenation. This study investigates the effects of both acute and short-term oral supplementation of Shoden (Ashwagandha extract) intake on performance and rate of perceived exertion in high-intensity aerobic and anaerobic exercise.

DETAILED DESCRIPTION:
Only a few clinical trials have looked at the effects of Ashwagandha in exercise and training. The studies had a dosage of 2 x 300 mg & 2 x 500 mg per day for 8 weeks and found to stimulate effects of strength training on muscle strength and muscle mass (Wankhede et al., 2015) and small increments in time to exhaustion and VO2max (Shenoy et al., 2012). However, the training intervention in both the studies were not adequately controlled and did not make a distinction between the acute and short-term effects of Ashwagandha intake.

Moreover, a lot of herbal supplements are commercially available containing majority of alkaloids and small amount of withaferine. European Food Safety Authority (EFSA) has categorized anaferine, anahygrine, withanine, sominiferine, somnine, tropine etc as toxic and harmful. Apart from alkaloids, withaferine A has also been categorized as cytotoxic lactones by EFSA. The Ashwagandha extract developed by Arjuna Natural Ltd is free from these alkaloids and is standardized to contain about 35% glycowithanolides.

This study will be a randomized, double blinded, placebo controlled, two treatment, crossover study and will be conducted in 2 phases ( acute & short term) with a total of 5 identical test sessions. Each test session involves a maximal incremental cycling test followed by a 90-sec maximal cycling performance test (day 1), and a 30-min simulated time-triaI on a cycling ergometer (day 2). Day 1 and day 2 are separated by a 24hr rest interval and for each subject it will be consistently scheduled on the same time of the day in order to eliminate a potential impact of diurnal variation in the results.

ELIGIBILITY:
Inclusion Criteria:

* Males between 18 and 35 years old
* Physically fit and involved in physical fitness training, or in individual or team sport activity for 2-4hours per week, or 3-6 hours per week for cycling
* Body mass index between 18 and 25
* Good health status confirmed by a medical screening

Exclusion Criteria:

* Any kind of injury/pathology that is a contra-indication to perform high-intensity exercise.
* Intake of any medication or nutritional supplement that is proven to affect exercise performance
* Intake of analgetics, anti-oxidants, or anti-inflammatory agents from 2 weeks prior to the start of the study
* More than 3 alcoholic beverages per day, including a maximum of one glass of wine per day
* Blood donation within 3 months prior to the start of the study
* Smoking
* Involvement in elite athletic training at a semi-professional or professional level
* Current participation in another research trial
* Any other argument to believe that the subject is unlikely to successfully complete the full study protocol

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Physically fit and involved in physical fitness training, or in individual or team sport activity for 2-4hours per week, or 3-6 hours per week for cycling
Enrollment: 12 (Estimated)
Dates: Start 2018-08-06 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Performance (mean power output (Watt)) | 30-min simulated time trials
  Simulated time trial on cycling ergometer (Avantronic Cyclus2)

SECONDARY OUTCOMES:
Rate of perceived exertion | At the end of incremental VO2 max test ; halfway (15 min) and at the end (30 min) of the 30 min time trial; on cycling ergometer
  15-point Borg rating scale of perceived exertion (ranging from 6 to 20, where 6 means "no exertion at all",13-14 means "somewhat hard" and 20 means "maximal exertion".). A number is chosen from the scale by an individual that best describes their level of exertion during physical activity.
Capillary Lactate | Incremental VO2 max test - middle and at the end of each incremental step ; 90s VO2 max test - just before the start of the test and 4 min following exhaustion; 30-Min Time Trial - 5-min intervals
  Blood samples from earlobes (Lactate Pro1, Arkray, Japan)
Oxygen Intake (VO2Max) | Measured during Incremental, 90s, and 30 min time trial.
  Highest oxygen uptake rate measured over a 30-s time-interval at the end of the test.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Hespel, Prof, Principal Investigator — Department of Kinesiology - KU Leuven
Locations (1):
- KU Leuven Athletic Performance Center / Bakala Academy, Leuven, Heverlee, Belgium

IPD SHARING:
Plan to Share IPD: Undecided
Data sharing can be carried out through a proper research proposal to the scientific review board of Arjuna Natural Ltd except in cases where Arjuna Natural Ltd. has no legal authority because the product has been out-licensed to another company or there is no feasible means to anonymise the data and redact personally identifiable information without compromising the privacy and confidentiality of research participants.